CLINICAL TRIAL: NCT05660577
Title: A Study to Evaluate the Product Performance of a New Silicone Hydrogel Multifocal Contact Lens
Brief Title: Evaluation of Product Performance of a New Silicone Hydrogel Multifocal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL916
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-02

CONDITIONS: Myopia and Hyperopia and Presbyopia
MeSH Terms: conditions — Myopia; Hyperopia; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- e Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens (Experimental)
  Interventions: Device: new silicone hydrogel daily disposable multifocal contact lens, the Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens

INTERVENTIONS:
Device: new silicone hydrogel daily disposable multifocal contact lens, the Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens — new silicone hydrogel daily disposable multifocal contact lens, the Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens

SUMMARY:
The objective of this study is to evaluate the product performance of a new silicone hydrogel daily disposable multifocal contact lens, the Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens, when worn by current soft contact lens wearers on a daily disposable wear basis

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 40 years or older on the date the ICF is signed and have the capacity to provide voluntary informed consent
* Subjects must be willing and able to comply with all treatment and follow-up/study procedures, as well as willing and able to refrain from using any contact lenses other than those provided for the duration of the study
* Subjects must be correctable through spherocylindrical refraction to 42 letters (0.1 logMAR) or better (distance, high contrast) in each eye
* Subjects must have clear central corneas and be free of any anterior segment disorders
* Subject must wear their current lenses for a minimum of 12 hours per day at least four days per week
* Subjects must habitually wear a multifocal lens in each eye
* Subjects must be an adapted multifocal soft contact lens wearer for a minimum of 6 months
* Subjects must require distance lens correction from +3.00 to -6.00 D in each eye
* Subjects must be presbyopic and require near add correction from +0.75 to +2.50 D in each eye
* Subjects must have access to an internet connection to complete an online survey and be able to receive text message

Exclusion Criteria:

* Subjects participating in any drug or device clinical investigation within 30 days prior to entry into this study and/or plan to do so during the period of study participation
* Subjects who are women of childbearing potential (those who are not surgically sterilized or postmenopausal) are excluded from participation in the investigation if they meet any one of the following conditions:

  * She is currently pregnant
  * She plans to become pregnant during the study
  * She is breastfeeding
* Subjects with any systemic disease currently affecting ocular health or that, in the Investigator's opinion, may have an effect on ocular health during the course of the study
* Subjects with an active ocular disease
* Subjects who have had any corneal surgery (e.g., refractive surgery)
* Subjects who have worn gas-permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last 3 months
* Subjects who currently wear monovision or toric contact lenses
* Subjects who are not correctable to 32 letters (0.3 logMAR) with bilateral soft multifocal contact lenses
* Subjects with an ocular astigmatism >1.00 D in either eye
* Subjects with anisometropia (spherical equivalent) >2.00 D
* Subjects with any Grade ≥2 finding during the slit lamp examination. Subjects with corneal infiltrates of ANY GRADE are not eligible
* Any "Present" finding during the slit lamp examination that, in the Investigator's opinion, interferes with contact lens wear
* Any scar or neovascularization within the central 6 mm of the cornea. Subjects with minor peripheral corneal scarring (that does not extend into the central area) that, in the Investigator's opinion, does not interfere with contact lens wear are eligible for this study
* Subjects who are amblyopic
* Subjects using any systemic or topical ocular medication that will, in the Investigator's opinion, affect ocular physiology or lens performance
* Subjects who are allergic to any component in the study care products

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Eric White OD Inc, San Diego, California
  - Lee & Woo Optometry, San Francisco, California
  - Chester T Roe III MD Prof LLC, Denver, Colorado
  - Pearle Vision, Jacksonville, Florida
  - Eola Eyes, Orlando, Florida
  - Vision Health Institute, Orlando, Florida
  - Golden Vision, Sarasota, Florida
  - The Eyecare Studio, LLC, Decatur, Georgia
  - Family Eyecare Center, Leavenworth, Kansas
  - Kannarr EyeCare, Pittsburg, Kansas
  - Casco Bay EyeCare, Portland, Maine
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - Koetting Associates, St Louis, Missouri
  - Spectrum Eyecare, Jamestown, New York
  - Saccco Eye Group, Vestal, New York
  - Oculus Research, Raleigh, North Carolina
  - CORE, Inc., Shelby, North Carolina
  - West Bay Eye Associates, Warwick, Rhode Island
  - Total Eye Care, PA, Memphis, Tennessee
  - Optometric Physicians of Middle Tennessee, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | e Bausch + Lomb (Kalifilcon A) Daily Disposable Multifocal Contact Lens
Started | 301
Completed | 292
Not Completed | 9
Not completed — Discontinued | 9

BASELINE CHARACTERISTICS:
Groups:
- Bausch + Lomb (Kalifilcon A) Daily Disposable Multifocal Contact Lens: New silicone hydrogel daily disposable multifocal contact lens, the Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens: new silicone hydrogel daily disposable multifocal contact lens, the Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens
Arm/Group | Bausch + Lomb (Kalifilcon A) Daily Disposable Multifocal Contact Lens
Number analyzed (Participants) | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (6.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 252
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 294

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Agreeing With the Statement "Clear Vision: Near, Far, and In-between
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Bausch + Lomb (Kalifilcon A) Daily Disposable Multifocal Contact Lens: New silicone hydrogel daily disposable multifocal contact lens, the Bausch + Lomb (kalifilcon A) Daily Disposable Multifocal Contact Lens
Arm/Group | Bausch + Lomb (Kalifilcon A) Daily Disposable Multifocal Contact Lens
Number analyzed (Participants) | 294
Participants | 241

ADVERSE EVENTS:
Time Frame: 3-Week
Description: Ocular Adverse Events
Arm/Group | Bausch + Lomb (Kalifilcon A) Daily Disposable Multifocal Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/294
Serious Adverse Events (participants affected / at risk) | 0/294
Other Adverse Events (participants affected / at risk) | 0/294

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT05660577/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT05660577/SAP_001.pdf